CLINICAL TRIAL: NCT06057350
Title: Surgery Versus Endoscopic Resection for Incompletely Removed Early Colon CAnceR (SCAR)- a Randomized Controlled Trial
Brief Title: Surgery Versus Endoscopic Resection for Incompletely Removed Early Colon CAnceR
Acronym: SCAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Collaborators: Hôpital Edouard Herriot (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Nuovo Regina Margherita Hospital (Other); Karolinska Institutet (Other); Humanitas Clinical and Research Center (Other); Medical University of Gdansk (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other); University Hospital of North Norway (Other); Helse Stavanger HF (Other Government); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Michael Bretthauer, Co-Principal Investigator, Norwegian Department of Health and Social Affairs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK KULMU-B 613856
Record Dates: First submitted 2023-08-12; First posted 2023-09-28 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Treatment Side Effects; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery (Active Comparator): Patients randomized to surgery are treated according to current guidelines with either open, laparoscopic or robotic surgical segmental bowel resection corresponding to lymphovascular drainage of the cancer.
  Interventions: Procedure: Tumor removal
- EFTR (Endoscopic Full-Thickness Resection) (Experimental): Patients randomised to EFTR are treated using devices approved for eFTR in the European Union and affiliated countries for the indication as applied in the trial. Before EFTR, the scar is identified and documented. The colonoscope is then removed, the EFTR device mounted, the colonoscope re-introduced, and eFTR performed.
  Interventions: Procedure: Tumor removal

INTERVENTIONS:
Procedure: Tumor removal — Removal of incompletely removed early-stage colon cancer

SUMMARY:
Randomized head-to-head comparison trial among patients who have undergone incomplete endoscopic resection of early colon cancer to evaluate the benefits, harms and burdens, as well as the ecological footprint and cost-effectiveness of endoscopic full thickness resection (eFTR), a minimally invasive endoscopic treatment with a colonoscope, as compared to standard-of-care surgery.

Co-primary endpoints are

* Rate of severe adverse events classified as grade III to V according to the Clavien Dindo classification within 30-days after study treatment
* CRC recurrence or sign of lymph nodes or distant metastases at 3 years after randomization comparing the two treatment groups (eFTR versus surgery).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 40 years or older with endoscopic removal (snare or forceps polypectomy; endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) with R1 (resection margin <0.1mm23,40) or Rx resection margins of colon cancer (location proximal to the rectum (12 cm or more from the anal verge))
* No contraindication for colon surgery as deemed by the multidisciplinary tumor board (MTB) at the participating centre
* Absence of the following histopathological tumor features: poor differentiation, lymphovascular invasion, tumor budding grade B2-B3.
* No sign of disease beyond stage T1N0M0 on standard-of-care computed tomography imaging of the thorax, abdomen and pelvis41 and clinical evaluation
* Identifiable resection site with colonoscopy, either by visualizing a previously administered tattoo or by identification of a scar in the correct colon segment
* No other tumors or polyps larger than 10 mm in diameter in the colorectum at time of randomization
* Complete colonoscopy with adequate quality of bowel preparation (Boston Bowel Preparation Scale score ≤2 in all colonic segments) and photo or video documentation of the appendiceal orifice or ileocecal valve.
* No colonic strictures or severe diverticulosis.
* No prior CRC
* No other malignant disease which is not deemed cured
* No confirmed or suspected genetic cancer syndrome (10 or more adenomas/serrated lesions, adenomatous or serrated polyposis syndrome; Lynch or Lynch-like syndrome)
* No inflammatory bowel disease
* Written informed consent provided by before enrolment

Exclusion Criteria:

* all who do not fulfill inclusion criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Severe adverse events | 30 days
  Rate of severe adverse events classified as grade III to V according to the Clavien Dindo classification within 30-days after study treatment
CRC recurrence or sign of lymph nodes or distant metastases | 3 years
  Rate of CRC recurrence or sign of lymph nodes or distant metastases

SECONDARY OUTCOMES:
CRC recurrence or sign of lymph nodes or distant metastases at 1 year after study treatment | 1 year
  CRC recurrence or metastases
CRC recurrence or sign of lymph nodes or distant metastases at 5 years after study treatment | 5 years
  CRC recurrence or metastases
CRC survival and overall survival at 1,3 and 5 years after study treatment | 1, 3, 5 years
  CRC survival and overall survival
Rate of severe adverse events classified as grade III to V according to the Clavien Dindo classification within 1 year after study treatment | 1 year
  Severe adverse events
Rate of mild and moderate adverse events classified as grade I and II according to the Clavien Dindo classification at 30 days after study treatment | 30 days
  mild and moderate adverse events
Length of hospital stay after study treatment | 30 days
  Hospital stay
Hospital readmission rate after discharge within 30 days after study treatment | 30 days
  Hospital readmission
Technical success of the trial procedures, defined as completion of eFTR and surgery as planned with endoscopic complete en-bloc scar excision or complete surgical resection | 1 day
  Technical success
Duration of the study procedure | 1 day
  Duration of procedure
Environmental footprint of study procedures at 30 days after study treatment | 30 days
  Carbon dioxide emission in kgCo2 per procedure
Health related quality of life and functional outcomes after 30 days and one year | 30 days, 1 year
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (0-100 points; higher point scores mean higher QoL)

OTHER OUTCOMES:
Cost-effectiveness | 5 years
  Costs in dollars as compared to effectiveness

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (2):
  - Vestre Viken Hospital, Oslo, Akershus
  - Akershus University Hospital, Oslo
- Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No